CLINICAL TRIAL: NCT05747196
Title: The Safety and Feasibility of the eLym™ System for the Decongestion of Excess Lymphatic Fluid Via the Thoracic Duct in Acute Decompensated Heart Failure
Brief Title: The Safety and Feasibility of the eLym™ System
Acronym: DELTA-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: WhiteSwell, Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: DELTA-HF CIP-01
Record Dates: First submitted 2023-01-06; First posted 2023-02-28 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Heart; Decompensation, Congestive

STUDY DESIGN:
Intervention Model Description: The study protocol indicates that subjects signing consent will be "enrolled"; however, the number of subjects treated with the investigational device will be less due to screening for inclusion / exclusion criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Label Treatment Arm (Experimental): Hospitalized patients with acute decompensated heart failure that meet eligibility criteria will have an eLym System temporarily placed via left internal jugular access. The eLym System will be in place for up to 60 hours.
  Interventions: Device: WhiteSwell eLym System

INTERVENTIONS:
Device: WhiteSwell eLym System — The WhiteSwell eLym™ System is designed to treat congestion in Acute Decompensated Heart Failure (ADHF) patients. The device comprises two endovascular components, a Catheter and a Sheath, that are used in combination with a Console. The device is designed to create a low-pressure zone at the Thoracic Duct Outflow which is located adjacent to the venous angle (junction of the left subclavian vein and left internal jugular vein). This low-pressure region facilitates movement of fluid (lymph) from the interstitial compartment through the lymphatic system and the Thoracic Duct and into the intravascular space, while removal of fluids from the intravascular space is enabled using diuretic therapy. The treatment duration will be up to 60 hours.

SUMMARY:
The goal of this feasibility study is to evaluated the safety and performance of the WhiteSwell eLym System in the treatment of fluid overload or congestion in adult patients with Acute Decompensated Heart Failure (ADHF). The main question[s] it aims to answer are:

* Acute device safety (30 days)
* Chronic device safety (31-180 days)
* Primary performance Outcomes (Technical success and patient treatment outcomes)

Participants who are hospitalized for ADHF will be screened for treatment with the eLym System. The System, placed in a heart catheterization laboratory, will be temporarily placed for up to 60 hours to treat congestion. The patient will be followed during the hospital stay through discharge and have follow-up assessments at 30-, 60-, 90- and 180-days.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Subject is admitted to the hospital with a primary diagnosis of Acute Decompensated Heart Failure (ADHF)
3. Subjects receiving intravenous (IV) diuretic for decompensated heart failure and demonstrating fluid overload. This includes peripheral edema ≥2+ (on a 0 to 4+ scale) and a minimum of 1 of the following:

   * Jugular venous distension ≥10 cm H20;
   * Pulmonary edema as determined by auscultation or imaging;
   * Hepatojugular reflux;
   * Paroxysmal nocturnal dyspnea or ≥ two-pillow orthopnea;
   * Dyspnea at rest with respiration rate ≥20 per minute.
4. Total DAILY diuretic dose prior to admission of ≥80mg Lasix or equivalent
5. Renal function parameters as measured by estimated glomerular filtration rate (eGFR) ≥20 ml/min/1.73m2
6. Subject must meet on one of the following criteria:

   * Subject has had a heart failure hospitalization or worsening of heart failure event requiring IV diuretic therapy (in hospital, emergency room, urgent care, or HF clinic) within the previous 6 months;
   * Renal function as measured by eGFR ≥20 and ≤45 ml/min/1.73m2;
   * At initial HF admission, <600 ml of urine output within 6 hours of initial IV bolus or urine sodium of <50 mmol/L at 1-2 hours after initial IV diuretic dose.
7. Elevated N-Terminal (NT) Pro B-type Natriuretic Peptide (BNP) or BNP:

   * NT Pro BNP >1000 pg/ml (>1500 for subjects with atrial fibrillation);
   * BNP >250 pg/ml (>375 for subjects with atrial fibrillation).
8. Albumin >2.5 g/dL
9. Subject must be able to have device placement procedure within 96 hours of presentation to the hospital and still be demonstrating fluid overload at the time of device placement
10. Subject willing and able to complete study assessments and agrees to comply with all follow-up evaluations
11. Subject has provided written informed consent

Exclusion Criteria:

1. Ultrasound Screening Assessment Exclusion:

   * Subjects' anatomy is not compatible with product dimensions as defined on the eLym system labelling
2. Subjects requiring intravenous vasoactive therapies (e.g., vasodilators, inodilators, inotropes), mechanical ventilation, MCS, or ultrafiltration
3. Subject has experienced a thromboembolic event [e.g., pulmonary embolism (PE), deep vein thrombosis (DVT), transient ischemic attack (TIA), or cerebrovascular events (CVA)] within the previous 6 months
4. Subject has contraindications to systemic anticoagulation
5. Subject currently on Dabigatran
6. Subject with International Normalized Ratio (INR) >2.2 not due to anticoagulation therapy, hypercoagulable state including heparin-induced thrombocytopenia, or on novel anticoagulants (NOACs) that cannot be held for a minimum of 24 hours prior to eLym System placement Note: If subject's INR is >2.2 at the screening and baseline assessment, it may be repeated to assess eligibility up to the time of the procedure.
7. Previous intracranial bleed unless there is documentation that the patient can safely use anticoagulation for 3 days
8. Gastrointestinal (GI) bleeding within 6 months requiring hospitalization and/or transfusion.
9. Recent major surgery within 30 days if the surgical would is judged to be associated with increased risk of bleeding.
10. Platelet count <75 10^3/μL
11. Inability to tolerate anticoagulation therapy for up to 3 days
12. Subject with systolic blood pressure <85 millimeters of mercury (mmHg) at time of enrollment
13. Subject has severe liver disease, liver fibrosis, or hempatorenal syndrome
14. Subject has evidence of active blood stream infection or pneumonia
15. Sustained malignant arrhythmias [e.g., ventricular tachycardia/fibrillation) in the last 90 days]
16. Subject with acute coronary syndrome (ACS) in the last 3 months
17. Subject with severe concomitant disease expected to prolong hospitalization or expected to cause death in ≤ 90 days
18. Subject with a rhythm management device implanted within the last 45 days (i.e., cardioverter/defibrillator, pacemaker, cardiac resynchronization device)
19. Subject is pregnant or lactating. Women of childbearing age who are not post-menopausal or not surgically sterile will need to demonstrate a negative urine or serum test.
20. Physician discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Acute safety as assessed by the rate of acute adjudicated device-, treatment-, and procedure-related Serious Adverse Events | Device placement skin puncture to 30 days post therapy
  The rate of acute device-, treatment-, and procedure-related Serious Adverse Events (SAE) as adjudicated by an independent Clinical Events Committee will be reported.
Chronic safety as assessed by the rate of chronic adjudicated device-, treatment-, and procedure-related Serious Adverse Events (SAE) | Day 31 out to 180 days post therapy
  The rate of chronic device-, treatment-, and procedure-related Serious Adverse Events (SAE) as adjudicated by an independent Clinical Events Committee will be reported.
Technical system performance as measured by the rate of procedures that demonstrate the user's ability to deploy, activate and remove the system. | Device placement procedure through eLym System therapy end (therapy lasting less than or equal to 72 hours)
  The system's technical performance will be assessed by evaluating the rate of procedures in which the user is able to deploy, activate and remove the system.
Acute response to therapy as evaluated by changes in the patients' body weight | Baseline (prior to eLym therapy), after eLym therapy (less than or equal to 72 hours after therapy initiation) and at discharge from the hospital (expected 3 - 10 days after hospital admission)
  Patients' acute response to therapy will be evaluated by assessing changes in body weight as measured in kilograms at baseline (prior to eLym therapy), after eLym therapy (less than or equal to 72 hours after therapy initiation) and at discharge from the hospital (expected 3 - 10 days after hospital admission). The change in weight will be expressed as an absolute change and percent change with an expected decrease corresponding to a treatment response.
Acute response to therapy as evaluated by changes in patients' net fluid loss or gain (milliliters) | Baseline (prior to eLym therapy), after eLym therapy (less than or equal to 72 hours after therapy initiation) and at discharge from the hospital (expected 3 - 10 days after hospital admission)
  Patients' acute response to therapy will be evaluated by assessing changes in patients' net fluid loss or gain based in total intake and output over 24 hours and expressed in milliliters at baseline (prior to eLym therapy), after eLym therapy (less than or equal to 72 hours after therapy initiation) and at discharge from the hospital (expected 3 - 10 days after hospital admission). An expected net fluid loss would correspond to a treatment response.
Acute response to therapy as evaluated by assessing changes in patients' renal function using estimated glomerular filtration rate (eGFR) | Baseline (prior to eLym therapy), after eLym therapy (less than or equal to 72 hours after therapy initiation), discharge from the hospital (expected 3 - 10 days after hospital admission), and at 30 day follow-up
  Patients' acute response to therapy will be evaluated by assessing changes in renal function as measured by estimated glomerular filtration rate (eGFR) (ml/min/1.73 (2)) using the Modification of Diet in Renal Disease (MDRD) calculation. Stable renal function would indicate a neutral response to therapy.
Acute response to therapy as evaluated by assessing changes in patients' renal function using laboratory parameter serum creatinine | Baseline (prior to eLym therapy), after eLym therapy (less than or equal to 72 hours after therapy initiation), discharge from the hospital (expected 3 - 10 days after hospital admission), and at 30 day follow-up
  Patients' acute response to therapy will be evaluated by assessing changes in renal function as measured by changes in serum creatinine (mg/dL). Stable renal function would indicate a neutral response to therapy.
Acute response to therapy as evaluated by the need for intensified heart failure therapy(ies) over the course of the hospitalization | Patient enrollment through hospital discharge (typically 3 - 10 days from admission to the hospital)
  Patients' acute response to therapy will be evaluated by assessing the need for intensified heart failure therapies indicating a worsening of the patient's condition, specifically evaluating the use of mechanical circulatory support, intravenous inotropes, or intravenous venodilators.
Acute response to therapy as evaluated by assessing Extra Vascular Lung Water (EVLW) measured by Sensible Medical's ReDS technology. | Baseline (pre eLym System therapy) and post eLym System therapy (less than or equal to 72 hours after the initiation of therapy)
  Patients' acute response to therapy will be evaluated by assessing Extra Vascular Lung Water (EVLW) as measured by Sensible Medical ReDS technology. The digital readout is provide as percent (%) with increasing numbers indicating a higher percentage of lung water and more congestion. Normal is consider to be less than 30%. Assessments will be made on seated patients prior to and just after the completion of therapy (less than or equal to 72 hours after the initiation of therapy).
Patient Quality of Life as evaluated by the Kansas City Quality of Life Questionnaire (KCCQ). | Baseline, Hospital discharge (typically 3- 10 days post hospital admission), 30-, 90-, and 180-days after hospital discharge.
  Changes in patients' quality of life will be assessed based on responses to the Kansas City Cardiomyopathy Questionnaire (KCCQ). The KCCQ is a 23-item self-administered questionnaire developed to independently measure the patient's perception of their health status, which includes heart failure symptoms, impact on physical and social function, and how their heart failure impacts their quality of life (QOL) within a 2-week recall period. All items are measured on a Likert scale with 5-7 response options. All KCCQ scores are scaled from 0 to 100 and frequently summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent. The scale will be administered at baseline, hospital discharge, and 30- 90- and 180- days post discharge.
Chronic response to therapy as evaluated by assessing changes in N Terminal-Pro Brain Natriuretic Peptide (NT-ProBNP) or Brain Natriuretic Peptide (BNP) biomarker levels | Baseline and 30-, 90-, and 180-days after hospital discharge
  Changes in N Terminal Pro Brain Natriuretic Peptide in picograms/milliliter (pg/ml) (NT-ProBNP) or Brain Naturiretic Peptide picograms/milliliter (pg/ml)(BNP) will assessed to evaluate the patient heart failure status at baseline, 30-, 90- and 180- days. NT-ProBNP or BNP increases are noted with increased patient congestion. A reduction in NT-ProBNP or BNP would indicate a patient improvement. Changes in NT-ProBNP or BNP will be expressed as an absolute change and a percent change from baseline.
Long term patient outcomes as evaluated by the time (days) to rehospitalization for acute decompensated heart failure | Hospital discharge through 180 days post hospital discharge
  Patients' need for rehospitalization for acute decompensated heart failure will be reported as observed starting at hospital discharge post therapy through the 180-day follow up window. An independent clinical events committee will adjudicate hospitalizations for heart failure relatedness.

CONTACTS AND LOCATIONS:
Overall Officials: William Abraham, MD, Study Director — Ohio State University
Locations (11):
- Georgia (3):
  - Israeli-Georgian Medical Research Clinical Helsicore, Tbilisi, Georgia
  - Tbilisi Heart and Vascular Center, Tbilisi, Georgia
  - Tbilisi Heart Centre, Tbilisi, Georgia
- Wroclaw University Hospital and Clinics, Wroclaw, Poland
- Spain (7):
  - Hospital Clinic de Barcelona, Barcelona, Spain
  - Germans Trias i Pujol Hospital, Badalona
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Clinico San Carlos, San Carlos
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Clínico de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Biegus J, Lindenfeld J, Felker GM, Bakris G, Jonas M, Lala A, Kereselidze Z, Khabeishvili G, Gogorishvili I, Nunez J, Bayes-Genis A, Ponikowski P, Abraham WT. Design and rationale of the eLym System for Decompensation of Excess Lymphatic Fluid via the Thoracic Duct in Acute Heart Failure (DELTA-HF). ESC Heart Fail. 2025 Jun;12(3):1719-1726. doi: 10.1002/ehf2.15192. Epub 2024 Dec 24. PMID 39716986